CLINICAL TRIAL: NCT01809899
Title: Risks and Outcomes of Enhanced Consent in Symptom-provocation Research
Brief Title: Enhanced Consent for Symptom Provocation Research
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Time and funding ran out prior to full recruitment
Sponsor: Georgetown University (Other)
Responsible Party: Principal Investigator, Mary Ann Dutton, PhD, Professor, Georgetown University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 4295-033
Record Dates: First submitted 2009-08-27; First posted 2013-03-13 (Estimated); Results first posted 2018-01-24 (Actual); Last update posted 2018-01-24 (Actual); Status verified 2017-06

CONDITIONS: Trauma
Keywords: Trauma; Abuse; Domestic Violence; Rape; Assault; MRI
MeSH Terms: conditions — Wounds and Injuries | interventions — Consent Forms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Enhanced Consent Procedure (Experimental): Participants in this group will receive an enhanced consent that will be an hour longer than usual.
  Interventions: Behavioral: Enhanced consent procedure
- Consent as Usual Procedure (Active Comparator): Participants in this group will receive a normal consent procedure to the study
  Interventions: Behavioral: Consent as Usual

INTERVENTIONS:
Behavioral: Enhanced consent procedure — Enhanced consent entails a more detailed consent procedure
  Arms: Enhanced Consent Procedure
Behavioral: Consent as Usual — Routine informed consent procedures
  Arms: Consent as Usual Procedure

SUMMARY:
The overall goal of the proposed study is to insure the protection and safety of human subjects who have been previously exposed to interpersonal traumatic events and who are participants in symptom provocation research. The investigators intend to examine trauma history, cognitive, interpersonal, and genetic predictors of participants' unfavorable reaction to participation in research involving trauma-related script-driven imagery (SDI). The design includes comparing participants in a consent as usual group to participants in an enhanced consent group to see which minimizes unfavorable effects of participating in a research provocation study. In addition, the two different consent groups will be assessed for their effects on psychobiological and neurobiological stress response. Furthermore, the investigators will examine the relationship between the psychobiological responses and neural mechanism during SDI, and unfavorable reactions to participation in symptom provocation research.

DETAILED DESCRIPTION:
The overall goal of the proposed study is to insure the protection and safety of human subjects who have been previously exposed to interpersonal traumatic events and who are participants in symptom provocation research. The investigators intend to examine trauma history, cognitive, interpersonal, and genetic predictors of participants' unfavorable reaction to participation in research involving trauma-related script-driven imagery (SDI). The design includes comparing participants with and without Posttraumatic Stress Disorder (PTSD) in a consent as usual group to participants in an enhanced consent group to see which group minimizes unfavorable effects of participating in a research provocation study. In addition, the two different consent groups will be assessed for their effects on psychobiological and neurobiological stress response. Furthermore, the investigators will examine the relationship between the psychobiological responses and neural mechanism during SDI, and unfavorable reactions to participation in symptom provocation research.

ELIGIBILITY:
Inclusion Criteria:

* nonsmoker
* female
* between 18-55
* experienced trauma
* willing to have a brain scan
* provide consent

Exclusion Criteria:

* alcohol abuse or dependence
* bipolar disorder
* suicidal intent
* metal in the body or anything else that would interfere with an MRI
* claustrophobia or inability to lie still for 45 minutes
* receiving current counseling
* on certain antidepressants, benzodiazepines, or other psychotropic medication
* pregnant or nursing

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2009-04; Primary Completion 2010-06 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary Ann Dutton, PhD, Principal Investigator — Georgetown University

IPD SHARING:
Plan to Share IPD: No
Data was not valid due to error in data collection technology

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 12 participants were recruited, but we were unsuccessful in recruiting sufficient number of non-PTSD, but trauma exposed patients.
Groups:
- Enhanced Consent Procedure: Enhanced consent includes use of teach back methods, video clips illustrating various study methods, and repeated confirmation of consent.
- Consent as Usual: Consent as Usual, with no Enhanced Consent features
Period: Overall Study
Arm/Group | Enhanced Consent Procedure | Consent as Usual
Started | 8 | 4
Completed | 8 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Enhanced Consent Procedure: Participants in this group will receive an enhanced consent that will be an hour longer than usual.
  Consent procedure: Enhanced consent entails a more detailed consent procedure than is routine.
- Total: Total of all reporting groups
Arm/Group | Enhanced Consent Procedure | Consent as Usual Procedure | Total
Number analyzed (Participants) | 8 | 4 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 4 | 12
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 4 | 12
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 8 | 4 | 12

OUTCOME MEASURES:

1. Primary Outcome: Blood Oxygen-Level Dependent (BOLD) Signal
Description: Functional Magnetic Resonance Imaging (fMRI). We were examining differences in Blood Oxygen-Level Dependent (BOLD) signal indicating reaction to a stress-provocation paradigm between the Enhanced Consent and Consent as Usual conditions.
Time Frame: Baseline
Population: No analyses were conducted due to an error in the scanner that resulted in no usable neuroimaging or physiological data. This includes the BOLD signal as well as the heart rate data and all other data collected while in the scanner.
Groups:
- Enhanced Consent Procedure: Enhanced Consent Procedure involved enhanced Institutional Review Board (IRB) consent procedures.
- Consent as Usual: Consent as Usual, involving no Enhanced Consent features
Arm/Group | Enhanced Consent Procedure | Consent as Usual
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Heart Rate
Description: Heart rate was measured while in the scanner as a secondary psychobiological outcome to be considered in tandem with the BOLD signals from the scanner.
Time Frame: Baseline
Population: as for outcome 1
Groups:
- Enhanced Consent Procedure: Enhanced Consent Procedure involved enhanced IRB consent procedures.
Arm/Group | Enhanced Consent Procedure | Consent as Usual
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Groups:
- Enhanced Consent Procedure: Participants in this group will receive an enhanced consent that will be an hour longer than usual.
  Consent procedure: Enhanced consent entails a more detailed consent procedure
- Consent as Usual Procedure: Participants in this group will receive a normal consent procedure to the study
  Consent procedure: Enhanced consent entails a more detailed consent procedure
Arm/Group | Enhanced Consent Procedure | Consent as Usual Procedure
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/4
Other Adverse Events (participants affected / at risk) | 0/8 | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes